CLINICAL TRIAL: NCT03630718
Title: Randomized Controlled Trial of Psychoeducational and Hypnosis Interventions on the Fatigue Associated With Primary Biliary Cholangitis in Women (CBP-HOPE)
Brief Title: Trial of Psychoeducational and Hypnosis Interventions on the Fatigue Associated With PBC in Women
Acronym: CBP-HOPE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: University of Paris 5 - Rene Descartes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: K180401J
Record Dates: First submitted 2018-06-15; First posted 2018-08-15 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Liver Cirrhosis, Biliary
Keywords: Liver Cirrhosis, Biliary; Female; Cholangitis; Hypnosis; Psychological treatment
MeSH Terms: conditions — Liver Cirrhosis, Biliary; Cholangitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control Group (CG) (No Intervention): Patients assigned to no intervention
- Psychoeducational Intervention Group (EG-EDU) (Active Comparator): Patients assigned to psychoeducational intervention
  Interventions: Behavioral: Psychoeducational Intervention
- Hypnosis intervention Group (EG-HYP) (Active Comparator): Patients assigned to hypnosis intervention
  Interventions: Behavioral: Hypnosis intervention

INTERVENTIONS:
Behavioral: Psychoeducational Intervention — The psychoeducational intervention will be a structured education programme and will consist of informing patients about fatigue dimensions, aetiology and treatments, by helping them to develop strategies to cope with fatigue better and by teaching them to manage the balance between activities and rest.
  The construction of the contents of the sessions of this intervention will aim to reduce fatigue via the programme developed by Reif et al. in cancer patients and is composed of 6 sessions of 90 minutes, one session per week. It is a group intervention for 8 patients. For this project, the investigators have reorganised the sessions and their content to fit with an individual format adapted to PBC. This format is more appropriate to take into account the specificity of the manifestation of fatigue for each patient.
  Other Names: EG-EDU
  Arms: Psychoeducational Intervention Group (EG-EDU)
Behavioral: Hypnosis intervention — The hypnosis intervention will consist of decreasing fatigue and the related distress, and increasing feelings of energy and well-being.
  Therefore, each hypnosis exercise will be audiotaped and given to the patient at the end of the session. Patients will be asked to use these recordings as much as they want to help them to manage fatigue. The techniques used are inspired by those used in chronic pain management and fatigue.
  Other Names: EG-HYP
  Arms: Hypnosis intervention Group (EG-HYP)

SUMMARY:
Fatigue is a clinical symptom that has been described as the most disturbing by around 50% of patients with PBC. It has an important impact on patients' quality of life and is associated with an increased mortality risk. To treat fatigue in PBC, only medical treatments have been tested with limited efficacy or serious sides' effects. In other diseases, mostly cancer, psychological interventions showed efficacy on fatigue decrease. Most interventions consist in psychoeducation with: education about fatigue, development of self-care or coping techniques, activity management and learning to balance between activities and rest. Hypnosis, which consists in a body work for psycho-therapeutic use (e.g., through imagination), has also shown promising results. Moreover, psychological intervention efficacy seems to be influenced by patients' characteristics, such as personality. Therefore, the first aim of the present single-center randomized controlled phase 2 trial is to assess the efficacy of a psycho educational intervention and a hypnosis intervention on PBC patients' fatigue to demonstrate that both psychoeducational and hypnosis interventions decrease patient fatigue.

ELIGIBILITY:
Inclusion Criteria:

* Women from 18 to 75 years old,
* Diagnosis of primary biliary cholangitis (PBC) according to recognized criteria (EASL 2017),
* Medically stable under treatment with UDCA initiated for at least 6 months, ie medically stable on the basis of liver biological parameters (no increase of more than 20% in bilirubin, ALP and transaminases) and absence of disabling pruritus (permanent and EVA> 6/10 or scratching lesions),
* Presenting a significant level of fatigue (fatigue score on PBC-40>= 33),
* Understanding the French language,
* Availability and ability of the patient to access an internet network terminal to answer the online questionnaires of the study,
* Signed consent form.

Exclusion Criteria:

* Presence of cirrhosis with a Child-Pugh B or C,
* Presence of disabling pruritus (permanent, or EVA>= 7/10 in the last 3 weeks, or objectivable scratching skin lesions),
* Patient on liver transplantation waiting list or total bilirubin> 50 μmol / L (3 mg / dL), or recent complication (<6 months) of cirrhosis (ascites, hepatic encephalopathy, rupture bleeding) of esophageal varices),
* Untreated depressive disorder,
* Any comorbidity not medically controlled (i.e. all dosage changes <3 months due to a control of the associated pathology deemed insufficient by the referring physician) or life-threatening in the medium term (within 2 years).
* Psychiatric disorder modifying the relationship to the reality

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2019-05-27 (Actual); Primary Completion 2023-05-17 (Actual); Study Completion 2023-05-22 (Actual)

PRIMARY OUTCOMES:
PBC-40 questionaire | At month 3

SECONDARY OUTCOMES:
Short Form Health Survey (SF36) (1) | At Day 0
Short Form Health Survey (SF36) (2) | At week 5
Short Form Health Survey (SF36) (3) | At month 3
Short Form Health Survey (SF36) (4) | At month 6
Multidimensional fatigue inventory (MFI) (1) | At Day 0
Multidimensional fatigue inventory (MFI) (2) | At week 5
Multidimensional fatigue inventory (MFI) (3) | At month 3
Multidimensional fatigue inventory (MFI) (4) | At month 6
PBC-40 questionaire (1) | At Day 0
PBC-40 questionaire (2) | At week 5
PBC-40 questionaire (3) | At month 6
Pittsburg Sleep Quality Inventory (PSQI) (1) | At Day 0
Pittsburg Sleep Quality Inventory (PSQI) (2) | At week 5
Pittsburg Sleep Quality Inventory (PSQI) (3) | At month 3
Pittsburg Sleep Quality Inventory (PSQI) (4) | At month 6
Epworth Sleeping Scale (ESS) (1) | At Day 0
Epworth Sleeping Scale (ESS) (2) | At week 5
Epworth Sleeping Scale (ESS) (3) | At month 3
Epworth Sleeping Scale (ESS) (4) | At month 6
Hospital Anxiety and Depression Scale (HADS) (1) | At Day 0
Hospital Anxiety and Depression Scale (HADS) (2) | At week 5
Hospital Anxiety and Depression Scale (HADS) (3) | At month 3
Hospital Anxiety and Depression Scale (HADS) (4) | At month 6

CONTACTS AND LOCATIONS:
Overall Officials: Christophe CORPECHOT, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Service hépatologie Hôpital Saint-Antoine, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Untas A, Goffette C, Flahault C, Vioulac C, Chazouilleres O, Soret PA, Ben Belkacem K, Gaouar F, Bernard N, Rousseau A, Corpechot C. PBC-HOPE: A Randomized Controlled Trial of Hypnosis and Psychoeducation in Women With Primary Biliary Cholangitis and Fatigue. Am J Gastroenterol. 2025 Jul 14. doi: 10.14309/ajg.0000000000003639. Online ahead of print. PMID 40658125